CLINICAL TRIAL: NCT06401239
Title: Investigating Dyadic Expectations About ARF Survivorship (IDEAS)
Acronym: IDEAS
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00429340; R01HL163660 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Failure; Caregiving Stress; Mental Health Issue
Keywords: ARF survivor; Caregiver; ICU recovery; Dyadic coping; Dyadic self-efficacy
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARF Survivor-Care Partner Dyads: The study will recruit 235 dyads of adult ARF survivors and care partners. The term "care partner" refers to an individual (e.g. family member or friend) that supports the survivor at home.
  Interventions: Other: Dyadic expectations about the ARF survivor's perceived health 6 months after hospital discharge; Other: Self-efficacy; Other: Concordant expectations/shared appraisal of ARF survivor's health 6 months after hospital discharge

INTERVENTIONS:
Other: Dyadic expectations about the ARF survivor's perceived health 6 months after hospital discharge — Dyad members' expectations will be collected at baseline and at 3- month follow-up assessments using a visual analogue scale (VAS) ranging from 0 - 100, similar to the EQ-5D-VAS.
Other: Self-efficacy — Self-efficacy in both dyad members will be assessed at 3- and 6-month follow-up assessments using the Generalized Self-Efficacy Scale (GSE). The GSE has 10 items scored on a 4-point scale. U.S. adult population norms are available.
Other: Concordant expectations/shared appraisal of ARF survivor's health 6 months after hospital discharge — Dyad members' expectations will be collected at baseline and at 3- month follow-up assessments using a visual analogue scale (VAS) ranging from 0 - 100, similar to the EQ-5D-VAS.

SUMMARY:
The purpose of this observational study is to understand how adults who survive acute respiratory failure (ARF) and the people (usually family) who support ARF survivors after returning home think about the first 6 months of recovery. The study aims to find out if expectations about the recovery process after ARF are associated with mental health symptoms in both survivors and the survivor's care partners. Study participants will complete 3 surveys over 6 months. These surveys ask questions about participants' future expectations, feelings, and mood. Surveys can be completed online, over the phone, or on paper.

DETAILED DESCRIPTION:
The overarching objectives of the Investigating Dyadic Expectations about ARF Survivorship (IDEAS) cohort study are to learn how expectations about ARF survivorship are related to dyadic mental health symptoms and dyadic coping. Specifically, the study aims are:

* Aim 1: To determine whether health expectations and self-efficacy after acute respiratory failure (ARF) are associated with mental health outcomes in survivor-care partner dyads.
* Aim 2: To assess whether concordant expectations within survivor-care partner dyads are associated with better dyadic coping (primary outcome) and exploratory secondary outcomes.

The term dyadic coping refers to the ways two people interact as the pair manage illness-related stressors. Concordant expectations within dyads, also called shared appraisal, refers to both members of a dyad being "on the same page", and is hypothesized to lead to better dyadic coping behaviors.

ELIGIBILITY:
Patient Inclusion Criteria:

* ≥18 years old
* Meets study definition of ARF:

  * The study defines ARF as meeting 1 of the following 3:

    1. Mechanical ventilation via an endotracheal tube ≥24 consecutive hours OR
    2. Non-invasive ventilation (CPAP, BiPAP) ≥24 consecutive hours that is not for obstructive sleep apnea or other stable use OR
    3. High flow nasal cannula with fraction of inspired oxygen (FIO2)≥.5 and flow rate ≥ litres per minute (LPM) for ≥24 consecutive hours.
  * Occasional rest periods of ≤1 hour are not deducted from the calculation of consecutive hours. Patients who are intubated for mental status or airway obstruction are not eligible unless they have simultaneous ARF.
* Survival to hospital discharge to home
* Speaks or reads English or Spanish
* Identifies an adult who is expected to act as a primary care partner for at least the next 6 months.

Patient Exclusion Criteria:

* Pre-existing cognitive impairment (IQ-CODE >3.6)
* Residing in a medical institution at hospital discharge
* Receiving hospice care or life expectancy <6 months
* Homelessness or recent history of psychosis

Care Partner Inclusion Criteria:

* ≥18 years old
* Speaks or reads English or Spanish

Care Partner Exclusion Criteria:

* Pre-existing cognitive impairment (IQ-CODE >3.6)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study team will enroll adults who were treated for ARF in ICUs at Johns Hopkins Hospital and Bayview Medical Center in Baltimore, Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Symptoms of Anxiety and Depression as Assessed by the Hospital Anxiety and Depression Scale (HADS) | 3 and 6 months after ARF survivor's ICU discharge
  Symptoms of anxiety and depression in both members of enrolled dyads will be assessed at 3- and 6-month follow-up assessments using the HADS. The HADS has 14 items. Scores for the anxiety and depression subscales range from 0 - 21 with scores ≥8 reflective of clinically significant symptoms.
Dyadic Coping as Assessed by the Dyadic Coping Inventory (DCI) | 3 and 6 months after ARF survivor's ICU discharge
  Dyadic coping will be assessed at 3- and 6-month assessments using the Dyadic Coping Inventory (DCI).The DCI contains 37 items that will be answered by both dyad members. Items are rated on a 5-point scale ranging from 1 ("Very rarely") to 5 ("Very often") and the total DCI score is the sum of items 1 through 35 after reverse coding negatively keyed items. There are established cut-off scores to evaluate dyadic coping as follows: DCI total score < 111 reflects below average dyadic coping, DCI between 111-145 reflects normal dyadic coping, and DCI total score > 145 reflects above average dyadic coping.

SECONDARY OUTCOMES:
Symptoms of Post Traumatic Stress as Measured by the Impact of Events Scale-Revised (IES-R) | 3 and 6 months after ARF survivor's hospital discharge
  Symptoms of Post Traumatic Stress in both members of enrolled dyads will be measured by the IES-R. The IES-R has 22-items, a total raw score range of 0-88, and subscales for Intrusion, Avoidance, and Hyperarousal. Higher scores indicate more symptoms of post-traumatic stress.
Health-related Quality of Life as Measured by the European Quality of Life 5-Domain 5-level Questionnaire (EQ-5D-5L) | 3 and 6 months after ARF survivor's hospital discharge
  The Health-related Quality of Life of the ARF survivor will be measured by the EQ-5D-5L. The EQ-5D-5L is made up of 6 items addressing mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and self-rated health. Index values will be calculated for the first 5 dimentions and converted to a US-based index value with negative values indicating states worse than death and 1.0 indicating perfect health. Self-rated health is assessed on a 0 - 100 scale with higher values indicating better perceived health. Population norms are available.
Social Isolation as Measured by Social Isolation Score | 3 and 6 months after ARF survivor's hospital discharge
  Social isolation experienced by both members of the enrolled dyad will be measured by a social isolation score developed by Pohl and colleagues for the National Health and Aging Trends Study (NHATS). The score is derived from responses to 5 questions and ranges from 0 to 6 with high scores indicating greater isolation.
Financial Toxicity as Assessed by Qualitative Questions | 3 and 6 months after ARF survivor's hospital discharge
  Financial Toxicity will be assessed by asking both members of the dyad whether the dyad have experienced 12 indicators of financial hardship since the index hospitalization. This list of indicators has previously been used in two peer-reviewed prospective cohort studies of people who survived hospitalization for COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Parker, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets and supporting information underlying publications will be shared at or prior to initial publication date.
Supporting Information: Study Protocol, Analytic Code
Time Frame: At or prior to publication dates.
Access Criteria: Datasets and associated metadata and documentation maintained by JHRDR is findable and identifiable through a digital object identifier (DOI) created by Johns Hopkins Data Services (JHRDR). Study data reposited in JHRDR will be available to the research community in perpetuity.

REFERENCES:
- [Background] Turnbull AE, Lee EM, Dinglas VD, Beesley S, Bose S, Banner-Goodspeed V, Hopkins RO, Jackson JC, Mir-Kasimov M, Sevin CM, Brown SM, Needham DM; Addressing Post-Intensive Care Syndrome-01 (APICS-01) Study Team. Health Expectations and Quality of Life After Acute Respiratory Failure: A Multicenter Prospective Cohort Study. Chest. 2023 Jul;164(1):114-123. doi: 10.1016/j.chest.2023.01.016. Epub 2023 Jan 19. PMID 36682611
- [Background] Vranceanu AM, Bannon S, Mace R, Lester E, Meyers E, Gates M, Popok P, Lin A, Salgueiro D, Tehan T, Macklin E, Rosand J. Feasibility and Efficacy of a Resiliency Intervention for the Prevention of Chronic Emotional Distress Among Survivor-Caregiver Dyads Admitted to the Neuroscience Intensive Care Unit: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2020807. doi: 10.1001/jamanetworkopen.2020.20807. PMID 33052404
- [Background] Geense WW, van den Boogaard M, van der Hoeven JG, Vermeulen H, Hannink G, Zegers M. Nonpharmacologic Interventions to Prevent or Mitigate Adverse Long-Term Outcomes Among ICU Survivors: A Systematic Review and Meta-Analysis. Crit Care Med. 2019 Nov;47(11):1607-1618. doi: 10.1097/CCM.0000000000003974. PMID 31464769
- [Background] Zante B, Camenisch SA, Schefold JC. Interventions in Post-Intensive Care Syndrome-Family: A Systematic Literature Review. Crit Care Med. 2020 Sep;48(9):e835-e840. doi: 10.1097/CCM.0000000000004450. PMID 32590386
- See also: Study description at NIH RePORTER — https://reporter.nih.gov/search/O7W6A0HPMkiJl6HuTKTxrw/project-details/10732929